CLINICAL TRIAL: NCT01661816
Title: Impact of Breast Cancer on Quality of Life of the Young Women, Her Life Partner and Her Couple
Brief Title: Breast Cancer and Quality of Life
Acronym: KALICOU
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: KALICOU
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; everyday issues; couple
MeSH Terms: conditions — Breast Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Within chemotherapy: 30 couples, interviewed within chemotherapy (6 to 8 months after diagnosis)
  Interventions: Behavioral: interview
- within Herceptin: 30 couples, within herceptin treatment (the first year after diagnosis)
  Interventions: Behavioral: interview
- within hormonotherapy: 30 couples, within hormonotherapy (between 2 and 7 years after diagnosis)
  Interventions: Behavioral: interview
- without hormonotherapy: 30 couples, did not received hormonotherapy (1 year after diagnosis)
  Interventions: Behavioral: interview
- end of treatment: 30 couples, after end of treatments for patients who did received hormonotherapy (7 years after diagnosis)
  Interventions: Behavioral: interview

INTERVENTIONS:
Behavioral: interview — psychological, emotional, family and social parameters

SUMMARY:
The study aims to analyse and decode interviews of patient with breast cancer, and then established according a multidimensional profile specific to the population and to create a questionnaire tha will allow a practical and qualitative evaluation of the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age < 45
* non metastatic breast cancer
* at least 6 months of relationship

Exclusion Criteria:

* no life partner
* inclusion criteria failure

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patient with breast cancer, diagnosed before aged 45, having a life partner
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
quality of life at different time of medical follow up | 6 months after diagnosis, 1 year after diagnosis, between 2 and 7 years after diagnosis, 7 years past diagnosis
  interviews with couples at different time frame depending on which group they are in

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - François Baclesse Center, Caen
  - Oscar Lambret Center, Lille
  - Gustave Roussy Institut, Paris
  - Hospital, Valenciennes